CLINICAL TRIAL: NCT03711864
Title: Safety and Efficacy of IM21 Car-t Cells in Patients With Recurrent or Refractory BCMA Positive Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Lu Zhang, Attending doctor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YMCART201804
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM21 CAR-T cells (Experimental): IM21 CAR-T cells
  Interventions: Biological: IM21 CAR-T cells

INTERVENTIONS:
Biological: IM21 CAR-T cells — fludarabine and cyclophosphamide Two days before cell infusion,all patients will be treated with fludarabine and cyclophosphamide for 3 days
  Other Names: IM21

SUMMARY:
In patients with multiple myeloma with recurrent or refractory BCMA, CAR-T cell infusion was performed after screening, blood collection and pretreatment. Starting dose for 5 x 10^5 / kg, 1 x 10^6 doses sequentially. If dose-limiting toxicity is not observed in 3 patients in a dose group, the next dose group test can be performed; If more than 2/3 of patients (2 cases, included) in a dose group had DLT, dose-escalation was not performed. If 1 case of DLT (1/3) appears in the first 3 patients of a dose group, 3 patients need to be added to the dose group (at this time, there are 6 patients in the group).

DETAILED DESCRIPTION:
In patients with multiple myeloma with recurrent or refractory BCMA, CAR-T cell infusion was performed after screening, blood collection and pretreatment. Starting dose for 5 x 10^5 / kg, 1 x 10^6 doses sequentially. If dose-limiting toxicity is not observed in 3 patients in a dose group, the next dose group test can be performed; If more than 2/3 of patients (2 cases, included) in a dose group had DLT, dose-escalation was not performed. If 1 case of DLT (1/3) appears in the first 3 patients of a dose group, 3 patients need to be added to the dose group (at this time, there are 6 patients in the group). If DLT occurs in 1 of the 3 patients (with or without) or 2 of the 6 patients (with or without), no further dose escalation is allowed. Researchers and bidders to form drug safety monitoring committee (SRC), every dose group of subjects to complete the DLT observation period, after summarizing the security of this dose group, determine the test of the next dose, subjects such as draw up the highest dose group safety tolerance, SRC to decide whether to continue to increase the dose group of research, finally according to have obtained all the safety and efficacy of dose group information to determine the recommended dose (RP2D).Dose-limiting toxicity (DLT)

ELIGIBILITY:
Inclusion Criteria:

1. The patient had multiple myeloma (according to the updated IMWG diagnostic criteria)Active (symptomatic) myeloma
2. Refractory and recurrent multiple myeloma Refractory definition: 1) treated with at least second-line bortezomib or lenalidomide 2) determined by the clinician Definition of recurrence: refer to NCCN clinical guidelines for multiple myeloma (2016. V2), including recurrence after transplantation.
3. Age: 18 to 80 years old;
4. The expected survival time was more than 3 months;
5. ECoG score 0-2 (refer to Annex 2)
6. Hemoglobin (HB)≥80g/L; absolute neutrophil count (ANC)>1×10^9/L; platelet count(PLT)≥50×10^9/L.

Those who voluntarily participated in the experiment and signed informed consent.

Exclusion Criteria:

1. High risk organ involvement patients: tumor invasion of central nervous system, gastrointestinal tract,lung,pericardium,one of the major vessels;
2. Those who have graft-versus-host reaction and need to use immunosuppressants, or who have autoimmune diseases;
3. Chemotherapy or radiotherapy was used within 3 days before blood collection;
4. Patients who used systemic steroids within 5 days before blood collection (except those who have recently or are currently using inhaled steroids);
5. The patients who used drugs to stimulate the production of bone marrow hematopoietic cells within 5 days before the blood collection period;
6. Those who have previously used any gene therapy products;
7. History of epilepsy or other central nervous system diseases;
8. New York Heart Association (NYHA) grade III or above (refer to Annex 3) (for patients with heart disease, this assessment is required);
9. Creatinine > 1.5 times normal upper limit, ALT / AST>3 times normal upper limit or bilirubin >2 times normal upper limit;
10. Active hepatitis B or hepatitis C virus, HIV or other uncured active infections;
11. Pregnant or lactating women;
12. Those who suffer from other uncontrolled diseases are not suitable to join the study; Any situation that the researchers believe may increase the risk of subjects or interfere with the test results.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2019-02-25 (Actual); Primary Completion 2021-10-10 (Estimated); Study Completion 2021-12-20 (Estimated)

PRIMARY OUTCOMES:
Occurrence of study related adverse events | 2 years
  defined as >= Grade 3 signs/symptoms, laboratory toxicities, and clinical events) that are possibly, likely, or definitely related to study treatment Adverse events assessed according to NCI-CTCAE v4.0 criteria 2.

CONTACTS AND LOCATIONS:
Overall Officials: Daobin Zhou, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China